CLINICAL TRIAL: NCT00951210
Title: Phase I Study of Intramuscular (IM) Injections of Allogeneic PLX-PAD Cells for the Treatment of Critical Limb Ischemia. PLX-PAD Are Mesenchymal-Like Stromal Cells Derived From a Full Term Placenta.
Brief Title: Safety of Intramuscular Injections (IM) of Allogeneic PLX-PAD Cells for the Treatment of Critical Limb Ischemia (CLI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1202-2
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2011-11

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease; Critical Limb Ischemia
Keywords: Peripheral Artery Disease; Peripheral Vascular Disease; Critical limb ischemia; PAD; CLI
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLX-PAD low dose (Experimental): IM injection Single treatment; multiple injections
  Interventions: Biological: PLX-PAD
- PLX-PAD high dose (Experimental): IM injection Double treatment; multiple injections
  Interventions: Biological: PLX-PAD

INTERVENTIONS:
Biological: PLX-PAD — IM injection

SUMMARY:
The purpose of this study is to determine the safety of PLX-PAD, Intra-muscular injections for the treatment of CLI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of critical limb ischemia defined as persistent, recurring ischemic rest pain for at least two (2) weeks, and/or ulceration or gangrene of the foot or toe, with ABI < 0.6 or/and TBI < 0.4
2. Rutherford category 4-5
3. Non candidate for revascularization or endovascular intervention based on unfavorable vascular anatomy or significant co-morbid medical conditions as confirmed by vascular study (e.g., angiogram, MRA) obtained within 3 months prior screening visit and signed approval of vascular surgeon. The decision to classify the subject as a non-candidate will be made by the investigator and confirmed by an independent third party vascular surgeon who is not participating in the study.
4. In the opinion of the investigator, major amputation is not anticipated over a period of three (3) months.
5. Those diabetic subjects who are on optimal diabetes medication, with an HbA1c < 8%

Exclusion Criteria:

1. Uncontrolled hypertension (defined as diastolic blood pressure > 110 mmHg or systolic blood pressure > 180 mmHg during screening).
2. Wounds with severity greater than Grade 2 on the Wagner Scale
3. Life-threatening ventricular arrhythmia - except if an ICD is implanted - or unstable angina - characterized by increasingly frequent episodes with modest exertion or at rest, worsening severity, and prolonged.
4. ST segment elevation myocardial infarction and/or TIA/CVA within six (6) months prior to enrollment.Patients with severe congestive heart failure (i.e. NYHA Stage IV)
5. In the opinion of the investigator, the patient is unsuitable for cellular therapy.

Ages: 40 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Adverse events; Amputation incidence, Death incidence & Rehospitalization incidence | 3 months
Immunological reaction | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cardiology PC, Birmingham, Alabama
  - Duke University Medical Center, Durham, North Carolina